CLINICAL TRIAL: NCT06571695
Title: Long Head of the Biceps Subpectoral Tenodesis Anatomic vs. Traditional Tensioning Technique During Rotator Cuff Repair: A Randomized Prospective Trial
Brief Title: Restoring the Anatomic Tension Relationship of the Long Head of the Biceps During Tenodesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Dane Salazar, Vice Chair and Professor of Orthopaedic Surgery, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 212671
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Biceps Tendon Disorder; Tendinosis; Rotator Cuff Injuries
MeSH Terms: conditions — Tendinopathy; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Anatomic Long Head of Biceps Tensioning Treatment Group vs. Traditional Long Head of Biceps Tensioning Control Group
Who Masked: Participant
Masking Description: The design will be a single blinded format where the surgeon will be aware of what treatment the patient will receive (Control vs. Intervention). The patient will not be informed of what arm of treatment they were selected for.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomic Long Head of Biceps Tensioning Technique (Experimental): Patients that are randomized to the intervention group will undergo biceps tenodesis in a standardized, step-by-step protocol as outlined in a previously published and publicly available article.
  Interventions: Procedure: Anatomic Long Head of Biceps Tensioning Technique
- Traditional Long Head of Biceps Tensioning Technique (Active Comparator): The control group patient will undergo biceps tenotomy and tenodesis based on surgeon feel on appropriate tensioning of the tendon (Current practice).
  Of note, there is no universal method or gold standard on how the long head of the biceps should be tensioned during bicep tenodesis.
  Interventions: Procedure: Traditional Long Head of Biceps Tensioning Technique

INTERVENTIONS:
Procedure: Anatomic Long Head of Biceps Tensioning Technique — The standard mini-open subpectoral approach will be made. The myotendinous junction of the long head of the biceps tendon and its location within the intertubercular groove will be marked using electrocautery. The surgeon will then turn to the glenohumeral joint and perform the biceps tenotomy.The long head of the biceps tendon will be retrieved.The tendon is tagged with a running, locking number 2 fiberwire suture at the mid substance of the myotendinous junction using the previously made electrocautery marks to set the tension. The tendon is shortened. The sutures from the biceps are passed through the Arthrex cortical button.The pectoralis major tendon is retracted and 2 centimeters proximal to the distal insertion a unicortical bone tunnel is drilled in the bicipital groove with a 3.2 millimeter drill.The wound is irrigated and the biceps button is threaded into this tunnel and then flipped.The suture is tensioned, securing the biceps against the groove
  Arms: Anatomic Long Head of Biceps Tensioning Technique
Procedure: Traditional Long Head of Biceps Tensioning Technique — Diagnostic arthroscopic shoulder scope will occur to assess the long head of the biceps for tendinopathy. Tenotomy will occur at the junction of the supraglenoid tubercle with arthroscopic scissors. Subsequent tensioning and tenodesis will be based on surgeon's preference
  Arms: Traditional Long Head of Biceps Tensioning Technique

SUMMARY:
The goal of this clinical trial is to determine the clinical impact of restoring the anatomic-tension relationship of the long head of the biceps (LHB) when performing a biceps tenotomy and tenodesis. The main question it aims to answer is whether anatomic tensioning will improve functional outcome scores and decrease postoperative complications. The investigators hypothesize that through a standardized method of anatomically tensioning the LHB tendon during tenodesis, patient outcomes will improve. Researchers will compare these outcomes to a control group receiving the traditional tensioning technique. Participants will be randomized to either the anatomic tensioning treatment group or the traditional tensioning control group.

DETAILED DESCRIPTION:
The long head of the biceps can be a source of anterior shoulder pain that is primarily due to inflammation or instability of the long head of the biceps (LHB) tendon . Patients that fail non-operative management become candidates for biceps tenotomy and tenodesis. Currently, there is no universal protocol or gold standard for how the LHB tendon is tensioned. At the investigators' institution, the LHB is tensioned based on individual surgeon feel for the correct tensioning. The purpose of this study is to conduct a randomized, single-blinded prospective study comparing patients with the current regimen of bicep tensioning vs. utilizing a standardized method of anatomically tensioning the LHB tendon. The primary aim of assessing change in the American Shoulder and Elbow Surgeon (ASES) scores from baseline to post-surgery between the control and intervention groups will be assessed using a student's t-test. In addition, longitudinal mixed effects models will be used to estimate changes in ASES scores, over all time-points using a random effect for surgeon. Other relevant patient characteristics such as age, sex, and Charlson score will be included to explore the adjusted relationship of the intervention and outcomes over time. A secondary aim of this study is to collect specific measurements of the myotendinous junction of the LHB tendon to potentially establish if any characteristics predispose patients to developing pathology of the LHB tendon.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age undergoing arthroscopic shoulder surgery
* Operations that occur at Loyola University Medical Center (Maywood, IL), Loyola Ambulatory Surgery Center (Maywood, IL), or Gottlieb Memorial Hospital

Exclusion Criteria:

* Previous shoulder surgery involving the long head of the biceps tendon
* Younger than 18 years old
* Current pregnancy. As per standard protocol with all surgeries, a urine pregnancy test is performed prior to surgery. If positive, the surgery will be cancelled and the patient will be excluded from the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] David TS, Schildhorn JC. Arthroscopic suprapectoral tenodesis of the long head biceps: reproducing an anatomic length-tension relationship. Arthrosc Tech. 2012 Jul 21;1(1):e127-32. doi: 10.1016/j.eats.2012.05.004. Print 2012 Sep. PMID 23766967
- [Background] Denard PJ, Dai X, Hanypsiak BT, Burkhart SS. Anatomy of the biceps tendon: implications for restoring physiological length-tension relation during biceps tenodesis with interference screw fixation. Arthroscopy. 2012 Oct;28(10):1352-8. doi: 10.1016/j.arthro.2012.04.143. Epub 2012 Aug 24. PMID 22925883
- [Background] Hussain WM, Reddy D, Atanda A, Jones M, Schickendantz M, Terry MA. The longitudinal anatomy of the long head of the biceps tendon and implications on tenodesis. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1518-1523. doi: 10.1007/s00167-014-2909-5. Epub 2014 Feb 27. PMID 24573238
- [Background] Jarrett CD, McClelland WB Jr, Xerogeanes JW. Minimally invasive proximal biceps tenodesis: an anatomical study for optimal placement and safe surgical technique. J Shoulder Elbow Surg. 2011 Apr;20(3):477-80. doi: 10.1016/j.jse.2010.08.002. Epub 2010 Oct 12. PMID 20943419
- [Background] Lafrance R, Madsen W, Yaseen Z, Giordano B, Maloney M, Voloshin I. Relevant anatomic landmarks and measurements for biceps tenodesis. Am J Sports Med. 2013 Jun;41(6):1395-9. doi: 10.1177/0363546513482297. Epub 2013 Apr 5. PMID 23562807
- [Background] Tao MA, Calcei JG, Taylor SA. Biceps Tenodesis: Anatomic Tensioning. Arthrosc Tech. 2017 Jul 24;6(4):e1125-e1129. doi: 10.1016/j.eats.2017.03.033. eCollection 2017 Aug. PMID 29354407
- [Background] Wolf RS, Zheng N, Weichel D. Long head biceps tenotomy versus tenodesis: a cadaveric biomechanical analysis. Arthroscopy. 2005 Feb;21(2):182-5. doi: 10.1016/j.arthro.2004.10.014. PMID 15689867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2020 to December 2022, 204 consecutive patients from Loyola University Medical Center were initially assessed for eligibility. The first participant was enrolled in October 27, 2020 and the last participant was enrolled in December 6, 2022.
Pre-assignment Details: Of 204 enrolled participants, 167 met inclusion criteria and were randomized to treatment.
Groups:
- Traditional Long Head of Biceps Tensioning Technique: The control group patient will undergo biceps tenotomy and tenodesis based on surgeon feel on appropriate tensioning of the tendon (Current practice).
  Of note, there is no universal method or gold standard on how the long head of the biceps should be tensioned during bicep tenodesis.
  Traditional Long Head of Biceps Tensioning Technique: Diagnostic arthroscopic shoulder scope will occur to assess the long head of the biceps for tendinopathy. Tenotomy will occur at the junction of the supraglenoid tubercle with arthroscopic scissors. Subsequent tensioning and tenodesis will be based on surgeon's preference
Period: Overall Study
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Started | 80 | 87
Completed | 79 | 81
Not Completed | 1 | 6
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique | Total
Number analyzed (Participants) | 80 | 87 | 167
Age, Continuous [Mean (Full Range); unit: years] | 54.8 [23.1 to 79.2] | 56.2 [30.3 to 76.4] | 55.5 [23.1 to 79.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 44 | 49 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 16 | 22
  White | 59 | 49 | 108
  More than one race | 13 | 20 | 33
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 80 | 87 | 167
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.8 (6.3) | 30.9 (6.0) | 30.9 (6.1)
Rotator Cuff Anteroposterior Tear Size [Mean (Standard Deviation); unit: millimeters] | 11.3 (7.6) | 13.0 (8.2) | 12.2 (7.9)
Surgery Right Side Laterality [Count of Participants; unit: Participants] | 50 | 55 | 105
American Shoulder and Elbow Surgeons Score [Mean (Standard Deviation); unit: units on a scale] | 42.4 (21.6) | 37.5 (18.1) | 39.9 (20.0)
Visual Analog Scale Pain Score [Mean (Standard Deviation); unit: units on a scale] | 5.7 (2.8) | 6.1 (2.4) | 5.9 (2.6)
Active Forward Flexion [Mean (Standard Deviation); unit: degrees] | 138.9 (29.4) | 138.2 (26.1) | 138.5 (27.7)
Active External Rotation [Mean (Standard Deviation); unit: degrees] | 45.8 (13.4) | 47.0 (10.6) | 46.4 (12.1)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of American Shoulder and Elbow Surgeon (ASES) Score Between Treatment and Control Groups
Description: The ASES form was created by the Society of the American Shoulder and Elbow Surgeons to help standardize outcome measures by both combining a physician-rated and patient rated section. The total maximum score (and best outcome) is 100. Half of the score is weighted for pain and the other half for function. The final pain score is calculated by subtracting the visual analog scale from 10 and multiplying by 5. For the functional portion, each of the 10 separate questions are on a scale from 0 to 3. The functional portion total is then multiplied by 5/3 to make it a total of 50 points. In summary, 50 points come from the visual analog scale and the other 50 come from the functional portion, which equals a possible total of 100.
Time Frame: 6 weeks
Population: Intention to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 44 | 39
units on a scale | 47.1 (20.7) | 37.1 (17.1)

2. Primary Outcome: Comparison of American Shoulder and Elbow Surgeon (ASES) Score Between Treatment and Control Groups
Description: as for outcome 1
Time Frame: 3 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 44 | 46
units on a scale | 59.5 (22.8) | 58.3 (22.5)

3. Primary Outcome: Comparison of American Shoulder and Elbow Surgeon (ASES) Score Between Treatment and Control Groups
Description: as for outcome 1
Time Frame: 6 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 39 | 38
units on a scale | 68.2 (32.6) | 73.1 (19.9)

4. Primary Outcome: Comparison of American Shoulder and Elbow Surgeon (ASES) Score Between Treatment and Control Groups
Description: as for outcome 1
Time Frame: 1 year
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 42 | 39
units on a scale | 60.0 (39.0) | 76.1 (19.5)

5. Primary Outcome: Comparison of American Shoulder and Elbow Surgeon (ASES) Score Between Treatment and Control Groups
Description: as for outcome 1
Time Frame: 1.5 years
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 79 | 81
units on a scale | 78.3 (22.5) | 77.3 (22.9)

6. Secondary Outcome: Comparison of Visual Analog Scale (VAS) Pain Score Between Treatment and Control Groups
Description: The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain progression, or compare pain severity between patients with similar conditions. The score ranges from 0-10 with 0 being pain free and 10 being severe pain.
Time Frame: 6 weeks
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 29 | 38
units on a scale | 4.8 (2.7) | 5.1 (2.6)

7. Secondary Outcome: Comparison of Visual Analog Scale (VAS) Pain Score Between Treatment and Control Groups
Description: as for outcome 6
Time Frame: 3 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 29 | 40
units on a scale | 3.6 (2.6) | 4.1 (2.6)

8. Secondary Outcome: Comparison of Visual Analog Scale (VAS) Pain Score Between Treatment and Control Groups
Description: as for outcome 6
Time Frame: 6 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 27 | 37
units on a scale | 2.0 (2.8) | 2.5 (2.4)

9. Secondary Outcome: Comparison of Visual Analog Scale (VAS) Pain Score Between Treatment and Control Groups
Description: as for outcome 6
Time Frame: 1 year
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 30 | 36
units on a scale | 1.5 (2.6) | 2.3 (2.3)

10. Secondary Outcome: Comparison of Visual Analog Scale (VAS) Pain Score Between Treatment and Control Groups
Description: as for outcome 6
Time Frame: 1.5 years
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 62 | 50
units on a scale | 2.2 (2.7) | 2.9 (3.2)

11. Secondary Outcome: Comparison of Active Forward Flexion Between Treatment and Control Groups
Description: Active forward flexion of the shoulder measured from 0 to 180 degrees
Time Frame: 6 weeks
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 63 | 72
degrees | 107.0 (45.1) | 97.8 (42.6)

12. Secondary Outcome: Comparison of Active Forward Flexion Between Treatment and Control Groups
Description: Active forward flexion of the shoulder measured from 0 to 180 degrees
Time Frame: 3 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 66 | 76
degrees | 138.7 (28.7) | 138.9 (26.7)

13. Secondary Outcome: Comparison of Active Forward Flexion Between Treatment and Control Groups
Description: Active forward flexion of the shoulder measured from 0 to 180 degrees
Time Frame: 6 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 51 | 66
degrees | 149.3 (20.1) | 145.8 (21.8)

14. Secondary Outcome: Comparison of Active Forward Flexion Between Treatment and Control Groups
Description: Active forward flexion of the shoulder measured from 0 to 180 degrees
Time Frame: 1 year
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 16 | 21
degrees | 150.3 (10.7) | 139.0 (28.5)

15. Secondary Outcome: Comparison of Active External Rotation Between Treatment and Control Groups
Description: Active external rotation of the shoulder measured from 0 to 90 degrees
Time Frame: 6 weeks
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 59 | 69
degrees | 33.1 (16.7) | 31.7 (13.0)

16. Secondary Outcome: Comparison of Active External Rotation Between Treatment and Control Groups
Description: Active external rotation of the shoulder measured from 0 to 90 degrees
Time Frame: 3 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 64 | 74
degrees | 43.1 (11.1) | 42.5 (11.2)

17. Secondary Outcome: Comparison of Active External Rotation Between Treatment and Control Groups
Description: Active external rotation of the shoulder measured from 0 to 90 degrees
Time Frame: 6 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 44 | 60
degrees | 46.3 (8.5) | 45.5 (10.8)

18. Secondary Outcome: Comparison of Active External Rotation Between Treatment and Control Groups
Description: Active external rotation of the shoulder measured from 0 to 90 degrees
Time Frame: 1 year
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
Number analyzed (Participants) | 13 | 18
degrees | 45.4 (4.8) | 43.6 (13.7)

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Anatomic Long Head of Biceps Tensioning Technique | Traditional Long Head of Biceps Tensioning Technique
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/87
Other Adverse Events (participants affected / at risk) | 0/80 | 0/87

LIMITATIONS AND CAVEATS:
The rate of response to pain, functional outcomes, and range of motion was low at most of the follow-up timepoints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT06571695/Prot_SAP_ICF_000.pdf